CLINICAL TRIAL: NCT02701920
Title: HeartLight: Heart Rate Monitoring for Newborn Resuscitation
Acronym: HeartLight
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Heartlight Systems Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 15099
Record Dates: First submitted 2016-02-25; First posted 2016-03-08 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2016-09

CONDITIONS: Infant, Newborn, Diseases; Fetus or Neonate Affected by Cesarean Section; Infant, Premature, Diseases
Keywords: Premature Birth; Infant; Heart rate
MeSH Terms: conditions — Infant, Newborn, Diseases; Infant, Premature, Diseases; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- NICU infants and hat: Newborn infants of any gestation on the neonatal intensive care unit (NICU).
  Interventions: Device: HeartLight hat; Device: The HeartLight hat with in-built sensor
- NICU infants and sensor: Newborn infants of any gestation requiring heart rate monitoring on the neonatal intensive care unit.
  Interventions: Device: The HeartLight hat with in-built sensor; Device: HeartLight; Device: HeartLight device
- Newborns and surgical delivery: Well term newborn infants following birth by cesarean section.
  Interventions: Device: The HeartLight hat with in-built sensor; Device: HeartLight; Device: HeartLight device
- Newborns needing stabilisation: Newborn infants requiring resuscitation or stabilisation following birth.
  Interventions: Device: HeartLight; Device: HeartLight device
- Parental feedback: Parental feedback of babies recruited into HeartLight will be sought.
  Interventions: Other: parental feedback
- Healthcare provider feedback: Healthcare professionals caring for babies recruited into HeartLight will have their feedback on the device sought.
  Interventions: Other: healthcare provider feedback

INTERVENTIONS:
Device: HeartLight hat — HeartLight hat will be worn for up to 1 hour.
  Groups: NICU infants and hat
Device: The HeartLight hat with in-built sensor — The HeartLight hat with in-built sensor will be worn.
  Groups: NICU infants and hat; NICU infants and sensor; Newborns and surgical delivery
Device: HeartLight — Electronic stethoscope will be used to estimate heart rate with HeartLight sensor/hat
  Groups: NICU infants and sensor; Newborns and surgical delivery; Newborns needing stabilisation
Device: HeartLight device — HeartLight sensor/hat will be used with ECG/Pulse oximetry/electronic stethoscope
  Groups: NICU infants and sensor; Newborns and surgical delivery; Newborns needing stabilisation
Other: parental feedback — Questionnaire
  Groups: Parental feedback
Other: healthcare provider feedback — Questionnaire
  Groups: Healthcare provider feedback

SUMMARY:
This study will compare a newborn heart rate sensor (HeartLight) that is integrated into a hat with other common forms of heart rate monitoring such as electrocardiography (ECG), stethoscope and pulse oximetry (PO) in newborn babies. This will help to evaluate the new heart rate sensor's reliability and accuracy.

DETAILED DESCRIPTION:
Up to 10% of newborns require some form of resuscitation at birth. Heart rate (HR) is the most sensitive indicator of resuscitation efficacy. HR is most commonly estimated using a stethoscope. However, in simulation studies it has been shown that newborn healthcare providers estimate HR incorrectly in up to 1/3 of cases. Common techniques for monitoring heart rate such as electrocardiography (ECG) and pulse oximetry (PO) were not developed for resuscitation at birth.

ECG, an established and accurate method of monitoring HR, is rarely used in the delivery room for a number of reasons including difficulty ensuring adhesion to the skin (the baby is wet/covered in vernix) and skin damage in premature babies caused by stripping of the electrodes. Current ECG systems also require 3 electrodes to be positioned which can delay resuscitation further. The usual site for transmission PO is the foot or hand. However, in newborn babies, and particularly those requiring resuscitation when the HR is low, blood flow is reduced so physiological mechanisms preserve brain and heart blood flow at the expense of other less important organs and limbs. As a consequence of this and the choice of wavelengths, it can be more difficult to obtain a reliable HR from POs on the limbs, and they typically obtain an HR after 1-2 minutes.

In the delivery room, ECG and PO systems have a requirement for cables to connect to the main monitors. These can get in the way and it is now recommended for many babies to delay cutting the umbilical cord (to ensure more blood enters the baby from the placenta) which often requires the baby to be resuscitated very close to the mother and even between their legs.

The HeartLight system is a wireless optical sensor within a custom newborn hat to allow quick and accurate HR monitoring. It will be compared to ECG, PO and electronic stethoscope to determine the accuracy and reliability. The trial has 4 phases; Phase 1 evaluates the thermal properties of the hat, Phase 2 evaluates the accuracy and reliability of the HeartLight sensor on babies within the Neonatal Intensive Care Unit environment, Phase 3 evaluates the HeartLight sensor in newborn babies born by cesarean section and Phase 4 evaluates the performance of the HeartLight sensor in babies of all gestations requiring resuscitation and stabilisation at birth.

The investigators anticipate the HeartLight sensor and hat will allow swift and effective deployment, reduce delays in resuscitation (due to using a stethoscope) and improve HR accuracy (as a result of avoiding errors in the usual manual mental calculations made in the stressful environment of the delivery room) when it is needed most. However, an additional benefit is that it will not require significant modification to the existing care pathway or resuscitation protocols, and therefore a potential barrier to clinical uptake is removed.

ELIGIBILITY:
Inclusion Criteria:

* Written consent from the mother
* Realistic prospect of survival as determined by the attending clinical team

Phase 1:

- Infants on NICU

Phase 2:

- Infants on NICU requiring heart rate monitoring

Phase 3:

- Newborn infants following non-emergency elective cesarean section

Phase 4:

- Newborn infants who attending clinical team anticipate will require assessment of heart rate at time of birth

Feedback:

* Mothers of babies recruited into HeartLight study
* Healthcare professionals exposed to the new device

Exclusion Criteria:

Phase 1+2:

* Infants undergoing palliative care
* Infants too sick to tolerate additional procedures

Phase 3:

* Abnormal antenatal scans suggesting significant fetal abnormality (by definition these are not routine pregnancies).
* Any infant in whom resuscitation is likely to be required.
* If multiple births then only the first baby born shall be recruited (due to resource limitations with researchers attending the birth)

Phase 4:

* Infants <23 weeks
* Infants that are not for active resuscitation as decided by the clinical team
* If multiple births then only the first baby born shall be recruited (due to resource limitations with researchers attending the birth)

Feedback:

Unable to obtain written informed consent

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Heart Rate acquisition time in the first minute of life | 1 hour
  Time to acquire heart rate from new optical hat sensor from birth should be within 1 minute of birth.

SECONDARY OUTCOMES:
Reliability of heart rate generated by HeartLight device | 1 hour
  Assess the reliability of the new heart rate device
Accuracy of heart rate generated by HeartLight device | 1 hour
  Assess the accuracy of the new heart rate device
Feedback on acceptability of hat and device | 1 hour
  Feedback will be recorded via a questionnaire from both healthcare professionals and mothers.
Thermal imaging to determine heat loss whilst wearing hat | 1 hour
  Participants will be thermal imaged whilst wearing the hat to determine heat loss.
Thermal imaging to determine heat loss during stabilisation and/or resuscitation | 1 hour
  Participants will be thermal imaged during stabilisation and/or resuscitation whilst wearing the hat to determine heat loss.

CONTACTS AND LOCATIONS:
Overall Officials: Don Sharkey, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes